CLINICAL TRIAL: NCT05027087
Title: The Effect of a Novel Blueberry Supplement on Dry Eye Disease (PLUM)
Brief Title: The Effect of a Novel Blueberry Supplement on Dry Eye Disease
Acronym: PLUM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SightSage Foods and Nutrition Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 43221
Record Dates: First submitted 2021-08-25; First posted 2021-08-30 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants receive the blueberry gummy supplement
  Interventions: Dietary Supplement: Blueberry gummy
- Placebo (Placebo Comparator): Participant receive the placebo gummy supplement
  Interventions: Dietary Supplement: Placebo gummy

INTERVENTIONS:
Dietary Supplement: Blueberry gummy — Gummy bear containing blueberry powder
  Arms: Treatment
Dietary Supplement: Placebo gummy — Gummy bear with no active ingredients
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy of a novel oral supplement (gummy bear) with blueberry powder on reducing dry eye signs and symptoms and assess its safety.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

1. Is at least 18 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. Is willing and anticipates to be able to comply with the daily intake of 3 gummy bears twice daily for 4 weeks;
5. As per TFOS DEWS II13, has dry eye symptoms as determined by an OSDI score ≥ 13 OR DEQ-5 ≥ 6, and at least one of the following:

   1. Tear film osmolarity ≥ 308 mOsm/L or interocular difference > 8 mOsm/L
   2. Non-invasive tear film break-up time of <10 seconds in at least one eye
   3. More than 5 spots of corneal staining OR > 9 conjunctiva spots OR lid margin staining (≥ 2mm length & ≥ 25% width) in at least one eye.

Exclusion Criteria:

A person will be excluded from the study if he/she:

1. Is participating in any concurrent clinical or research study;
2. Currently wears, or has worn contact lenses in the past 3 months;
3. Has symptoms/ signs of severe dry eye, defined by an OSDI score ≥ 33 and at least one of the following:

   1. Corneal staining grade ≥ 3 (Oxford scale)
   2. Non-invasive tear film break-up time of ≤ 3 seconds in at least one eye;
4. Has any known active* ocular disease and/or infection;
5. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
6. Is using any systemic or topical medications (including topical corticosteroids/ NSAIDs or glaucoma medications) that in the opinion of the investigator may affect a study outcome variable;
7. Is currently taking, or has taken, any supplements containing anti-oxidants in the last three months;
8. Has started taking omega-3 supplements within the last 3 months or intend to start them during the study;
9. Has a known sensitivity or an allergy to ingredients of the gummy bears;
10. Has been diagnosed with glucose-6-phosphate dehydrogenase (G6PD) deficiency;
11. Has a known sensitivity to the diagnostic pharmaceuticals to be used in the study;
12. Is pregnant, lactating or planning a pregnancy at the time of enrolment (by self-report);
13. Has undergone refractive error surgery or intraocular surgery;
14. Is a member of CORE directly involved in the study;
15. Has taken part in another (pharmaceutical) research study within the last 30 days.

    * For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and mild dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Change in ODSI score from Baseline | 4 weeks
  The Ocular Surface Disease Index (OSDI) is a 12-question validated questionnaire used to measure ocular symptoms, visual function, and environmental factors that may affect a patient's vision. The OSDI scoring scale ranges from 0 to 100. The lower the score, the more symptomatic relief from dry eye symptoms a patient experiences. Change between the score at baseline and the score at 4 weeks is reported.
Change in Non-Invasive Tear Break-Up Time (NITBUT) from Baseline | 4 weeks
  The time required for a dry spot to appear on the corneal surface after blinking is referred to as the tear film break-up time. The change in this time (measured in seconds) between baseline and 4 weeks is reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Ocular Research & Education, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No